CLINICAL TRIAL: NCT06140329
Title: A Natural History Study in Patients With Genetically Confirmed Diagnosis of Autosomal Dominant Optic Atrophy (ADOA), Caused by OPA1 Mutation
Brief Title: Natural History of Autosomal Dominant Optic Atrophy (ADOA), Caused by OPA1 Mutation
Status: Terminated | Type: Observational
Why Stopped: The study was terminated due to low participant enrolment and to accommodate PYC's future interventional study.
Sponsor: PYC Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: PYC-001
Record Dates: First submitted 2023-11-15; First posted 2023-11-18 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Autosomal Dominant Optic Atrophy; Optic Atrophy, Autosomal Dominant; Optic Atrophies, Hereditary; Kjer Optic Atrophy
MeSH Terms: conditions — Optic Atrophy, Autosomal Dominant; Optic Atrophies, Hereditary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this study is to characterize the disease progression of confirmed OPA1 mutation-associated autosomal dominant optic atrophy (ADOA) by evaluating the changes in ocular structural and functional outcomes.

DETAILED DESCRIPTION:
This is a multi-center, longitudinal, prospective, observational natural history study of patients with confirmed OPA1 mutation (haploinsufficiency) associated ADOA. The study will be conducted at up to 10 sites across the United States, Australia and Europe.

Each participant's medical record will be reviewed for historical information, and clinical data will be recorded in a secure database. Natural history data will be collected prospectively and will include ophthalmic exams, imaging studies and electrophysiological testing. Assessments will be conducted as described in this protocol approximately every 3 months in the first year and every 6 months in the second year of the study after each participant's baseline visit

ELIGIBILITY:
Inclusion Criteria:

* Participants and/or their parent(s)/guardian(s) must have given written informed consent before any study-related activities are carried out and must be able to understand the full nature and purpose of the trial, including possible risks and adverse effects. Assent, where appropriate, will be obtained according to institutional guidelines.
* Males and females, 8 years of age and above.
* Have a clinical diagnosis of OPA1 mutation (haploinsufficiency) associated ADOA.
* No other ocular pathology.
* Patients with best-corrected visual acuity (BCVA) of between 20/40 (70 Early Treatment of Diabetic Retinopathy Study [ETDRS] letters) and 20/160 (39-43 ETDRS letters)
* Willing and able to comply with all study assessments and adhere to the protocol schedule and restrictions.
* For sites performing the Detection of apoptosis in retinal cells (DARC) procedure, and in volunteers ≥ 12 years only:

  1. Female volunteers must:

     I. Be of non-child-bearing potential at least 6 weeks before the screening visit or postmenopausal (where postmenopausal is defined as no menses for 12 months without an alternative medical cause), or

     II. If of childbearing potential, must:
     * Have a negative pregnancy test at the screening visit and prior to each administration of ANX776, and
     * Agree not to attempt to become pregnant or donate ova from signing the consent form until at least 30 days after the last dose of ANX776, and
     * Agree to use adequate contraception (defined as the use of a condom by the male partner combined with the use of a highly effective method of contraception from one month prior to screening until at least 30 days after the last dose of ANX776, if not exclusively in a same-sex relationship or abstinent as a committed lifestyle.
  2. Male volunteers must:

     * Agree not to donate sperm from signing the consent form until at least 90 days after the last dose of ANX776, and
     * If engaging in sexual intercourse with a female partner who could become pregnant, agree to use adequate contraception (defined as the use of a condom combined with the use of a highly effective method of contraception) from signing the consent form until at least 90 days after the last dose of study drug.

Exclusion Criteria:

* Participant has a known allergy to ANX776 or any of its excipients.
* Have any uncontrolled systemic disease that, in the opinion of the Investigator, would preclude participation in the study, which includes but is not limited to, infection, uncontrolled elevated blood pressure, cardiovascular disease, or glycemic control issues, or any other medical condition that may put the participant at risk due to study procedures. Note: comorbidities relevant to the pathogenesis of OPA1 associated ADOA (including hearing loss, peripheral neuropathy, myopathy, and ataxia) are acceptable.
* Have mutations in genes that cause ADOA, other than OPA1 (for example in case of dominant negative ADOA) and ADOA Plus.
* Within 3 months prior to Baseline (Visit 2), have undergone any vitreoretinal surgery (scleral buckle, pars plana vitrectomy, retrieval of a dropped nucleus or intraocular lens, radial optic neurotomy, sheathotomy, cyclodestructive procedures or multiple filtration surgeries [2 or more]) or any other ocular surgery.
* Have ocular media opacity or poor pupillary dilation prohibiting quality ophthalmic evaluation or photography, as assessed by the Investigator.
* Have used any investigational drug or device within 90 days or 5 estimated half-lives of Visit 2, whichever is longer, or plan to participate in another study of a drug or device during the study period. Participation in observational trials is allowable based on Investigator discretion and consultation with the Medical Monitor. It is assumed that the observational trial evaluations would not interfere with participation in this study.
* Have received any prior cell or gene therapy for a retinal condition.
* Have a recent history (<6 months) of or current excessive recreational drug or alcohol use, in the opinion of the Investigator. Note: excessive alcohol use is defined as regular consumption of > 10 standard drinks per week or > 4 standard drinks per day, where 1 standard drink is defined as 10 grams of pure alcohol.
* Any other condition or prior therapy that in the opinion of the Investigator would make the volunteer unsuitable for this study, including inability to cooperate fully with the requirements of the study protocol or likelihood of noncompliance with any study requirements.

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of approximately 40 participants (80 eyes) with a genetically confirmed OPA1 mutation.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2024-02-28 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-10 (Actual)

PRIMARY OUTCOMES:
Best-corrected High Contrast Visual Acuity (HCVA) | Baseline through Year 2
  Best-corrected high contrast visual acuity (HCVA) for both distance and near will be evaluated using the ETDRS electronic visual acuity charts and the MNRead acuity chart
Low Contrast Visual Acuity (LCVA) | Screening through Year 2
  Low contrast visual acuity (LCVA) for both distance and near will be evaluated using the low contrast ETDRS letter chart
Contrast Sensitivity | Baseline through Year 2
  Contrast sensitivity recorded using the Pelli-Robson chart
Color Vision | Baseline through Year 2
  Color vision tested using the Hardy Rand Rittler test
Retinal Thickness | Baseline through Year 2
  Change retinal thickness is measured using spectral domain optical coherence tomography (SD-OCT), as measured by the central reading center (SD-OCT), as measured by the central reading center
Ellipsoid Zone (EZ) Volume | Baseline through Year 2
  Change in EZ volume measured using spectral domain optical coherence tomography (SD-OCT), as measured by the central reading center
Ellipsoid Zone (EZ) Area | Baseline through Year 2
  Change in EZ area measured using spectral domain optical coherence tomography (SD-OCT), as measured by the central reading center
Visual Field Sensitivity | Baseline through Year 2
  Visual field sensitivity measured by automated static perimetry
Multifocal Visual Evoked Potential (mfVEP) | Baseline through Year 2
  The waveform of the evoked responses, the latency, and amplitude are analyzed.
Pregnancy Test | Baseline
  A urine human chorionic gonadotropin (hCG) pregnancy conducted in all women of childbearing potential (WOCBP) > 12 years of age at baseline. If a urine test is positive, the DARC procedure will not be performed.
DARC (Detection of Apoptosing Retinal Cells) | Baseline through Year 2
  The DARC test is conducted using an IV injection of fluorescently labelled Annexin V (called ANX776). Individual stressed and apoptotic retinal cells are visible as white spots on the image for DARC count, which are quantified using a confocal scanning laser ophthalmoscope using the indocyanine green angiography (ICGA) settings.
Flavoprotein Fluorescence (FPF) | Baseline through Year 2
  Functional imaging of mitochondria using Flavoprotein Fluorescence.
Retinal Abnormalities | Baseline through Year 2
  Ultrawide fundus photography is conducted OU to assess retinal abnormalities
Adverse Events (AEs) | Screening through Year 2
  Frequency of ocular adverse events (AEs)
Genomic Analysis for Study Eligibility | Screening
  OPA1 genetic testing at screening visit
Vital signs | Baseline through Year 2
  Vital signs assessments (pulse rate, body temperature, systolic and diastolic blood pressure, and respiratory rate) performed in participants undergoing the DARC assessment only.

SECONDARY OUTCOMES:
To determine the outcome measures that are associated with ADOA disease progression. | Baseline through Year 2
  To understand the disease progression in participants with confirmed OPA1 mutation-associated ADOA determined by changes in structural and functional markers from the primary outcome within the study period.

OTHER OUTCOMES:
To evaluate the safety of ANX776 in patients ≥ 12 years. | Baseline through Year 2
  Incidence, type and severity of treatment-emergent and treatment-related AEs in patients ≥ 12 years.
  Changes from baseline in vital signs (pulse rate, body temperature, systolic and diastolic blood pressure, and respiration rate) in patients ≥ 12 years.

CONTACTS AND LOCATIONS:
Overall Officials: Sreenivasu Mudumba, PhD, Study Chair — PYC Therapeutics
Locations (7):
- United States (2):
  - Bascom Palmer Eye Institute, Miami, Florida
  - University of Washington, Seattle, Washington
- Sydney Eye Hospital, Sydney, New South Wales, Australia
- Medical University of Graz, Graz, Styria, Austria
- CHU de Rennes, Rennes, Brittany Region, France
- Medizinische Hochschule Hannover, Hanover, Lower Saxony, Germany
- Amsterdam University Medical Centers, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No